CLINICAL TRIAL: NCT00220181
Title: A Prospective Study to Identify Changes in Nutritional Status and Bowel Symptoms in Patients Receiving a Course of Radical Radiotherapy to the Pelvis for Treatment of Gynaecological, Urological or Rectal Cancer.
Brief Title: Prospective Study in Pelvic Radiotherapy Patients
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Other Study IDs: CCR2240
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Gynaecological, Urological or Rectal Cancer
Keywords: Nutritional status; Bowel symptoms; Radical radiotherapy to pelvis; Gynaecological, urological or rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Symptoms such as diarrhoea and abdominal discomfort are common side effects of radiotherapy for tumours in the pelvis and usually occur within 2 weeks of starting treatment. Once the course of radiotherapy has been completed these symptoms usually subside, but in some patients they may continue and sometimes cause significant problems.

It is not clear what processes are occurring to trigger such symptoms. There are a number of possibilities and we would like to investigate these further. If we can identify specific reasons for symptoms being worse in one patient compared to another, then we can try to either prevent or treat these. The aim of this study is to look for differences in the way that the bowel adapts to radiotherapy in patients who do and those who don't experience bowel symptoms during their course of radiotherapy.

DETAILED DESCRIPTION:
Patients with pelvic cancers may be treated with radical radiotherapy as part of their disease management. Acute intestinal changes such as diarrhoea, abdominal pain and nausea ocur in about 75% of patients. Severe acute changes predispose to chronic, intractable intestinal changes. Nutritional intervention during radiotherapy may protect the bowel from toxicity.

A number of nutritionally related changes in bowel function may cause acute intestinal problems during radiotherapy. These include: Bile-acid & pancreatic enzyme potentiated damage to mucosa causing loss of epithelial integrity and in turn increased permeability to antigens and luminal bacteria; Bile-acid malabsorption, decreasing the gut's ability to digest fat; Reduced disaccharidase activity due to loss of the intestinal brush border, causing malabsorption of sugars leading to osmotic diarrhoea; Statis/ dysmotility in the small intestine prompting bacterial overgrowth.

There is little prospective data in patients undergoing radiotherapy to help to identify which are important. To understand what changes are relevant during a 6-week course of radiotherapy we plan this prospective observational study. Any changes identified in this study could be ameliorated by specific nutritional intervention in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with gynaecological, bladder or rectal malignancy about to embark ona 5-6 week course of radical radiotherapy to the pelvis who is able to give informed consent

Exclusion Criteria:

* Patients unable or unwilling to give informed consent
* Patients who have already started radiotherapy

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-04; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Jervoise Andreyev, Principal Investigator — Imperial College London